CLINICAL TRIAL: NCT01747005
Title: Effect of Enhanced Recovery After Surgery (ERAS) on Inflammatory Response After Planned Abdominal Hysterectomy: A Prospective Randomized Clinical Trial.
Brief Title: Effect of Enhanced Recovery After Surgery (ERAS) on Inflammatory Response After Planned Abdominal Hysterectomy
Acronym: GERAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Antypin Eduard Eduardovich (Other)
Collaborators: Northern State Medical University (Other)
Responsible Party: Sponsor-Investigator, Antypin Eduard Eduardovich, Anesthesiologist, Samoilova Maternity Home
Organization: Samoilova Maternity Home (Other)
Other Study IDs: SMH-0001
Record Dates: First submitted 2012-11-27; First posted 2012-12-11 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Hysterectomy
Keywords: abdominal hysterectomy; enhanced recovery after surgery; inflammatory response; ERAS; combined spinal-epidural anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum

GROUPS / COHORTS (2):
- Conventional therapy
- ERAS: Oral intake of solid food restriction 6 hours before surgery. Oral intake clear fluids restriction 2 hours before surgery. Intravenous 5% Dextrose-500 ml 1 hour before surgery. Intravenous dexamethasone -4mg before anesthesia. Combined spinal-epidural anesthesia. Intraoperatively 10 ml/kg intravenous of crystalloids. Paracetamol intravenous 1g. Early mobilization of patient. Oral solid food intake 4 hour postoperative. Postoperative continuous epidural analgesia.

SUMMARY:
The aim of study is to determine effect of enhanced recovery after surgery (ERAS) on inflammatory response after abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Abdominal hysterectomy
* ASA class I or II

Exclusion Criteria:

* psychiatric disorders
* ASA III and IV
* Chronic inflammatory disorders
* Pregnancy
* Local anesthetics allergy
* Coagulation disorders
* patients receiving anticoagulants

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted patients in maternity home
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change of Serum level of IL-1beta,IL-6,CRP,Cortisol,IL-4 by immuno-ferment analysis. | baseline, 24 hour post-operative and 7 days post-operative

SECONDARY OUTCOMES:
Change of postoperative pain, fatigue and postoperative nausea and vomiting | baseline,6,12,24,48 hour and 7 days postoperatively
  Postoperative pain will be assessed by visual analogue scale. Postoperative fatigue will be assessed by modified analogue scale. incidence of postoperative of nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Samoilova maternity home, Arkhangelsk, Arkhangelskya Oblast, Russia